CLINICAL TRIAL: NCT02006615
Title: The Role of Primary Motor Cortex and Prefrontal Cortex for Facilitation of Motor System and Working Memory in Stroke, Parkinson, and Elderly Patients
Brief Title: The Role of Primary Motor Cortex and Prefrontal Cortex for Facilitation of Motor System and Working Memory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal investigator, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-07-011A
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Central Nervous System Diseases
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High frequency rTMS plus fNIRS (Experimental): rTMS with neuroimage assessment of functional near infrared spectroscopy
  Interventions: Device: Functional near infrared spectroscopy; Device: rTMS
- Sham rTMS (Sham Comparator): Sham stimulation
  Interventions: Device: rTMS
- High frequency rTMS (Experimental): High frequency rTMS to modulate brain areas
  Interventions: Device: rTMS

INTERVENTIONS:
Device: Functional near infrared spectroscopy — Using high-sensitivity infrared to detect the active brain areas
  Other Names: fNIRS
  Arms: High frequency rTMS plus fNIRS
Device: rTMS — To modulate brain cortex

SUMMARY:
The investigators hypothesize that ten sessions of repetitive transcranial magnetic stimulation yield ability to upregulate the function of primary motor cortex and prefrontal cortex that play key roles in motor and frontal memory processing.

DETAILED DESCRIPTION:
Excitatory (>3Hz) rTMS could facilitate the brain cortex and neuroplasticity that benefits motor control and working memory when the coil is applied over primary motor cortex or dorsolateral prefrontal gyrus.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or hemorrhagic cerebrovascular lesion,
2. Parkinson's disease

Exclusion Criteria:

* Seizure
* With metal implantation
* Dementia or severe cognitive impairment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2021-07-11 (Estimated); Study Completion 2021-07-11 (Estimated)

PRIMARY OUTCOMES:
Change of Repeatable Battery for the Assessment of Neuropsychological Status | Up to 12 weeks
  Test cognition including memory, attention, language...

SECONDARY OUTCOMES:
Change of Montreal Cognitive Assessment | Up to 12 weeks
  Test cognition including memory, attention, and language.
Change of Fugl-Meyer Assessment , Wolf Motor Function Test | Up to 12 weeks
  Test upper limb motor function.

OTHER OUTCOMES:
Change of hand grip, pinch power | Up to 12 weeks
  Test hand strength.

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yi Tsai, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chang PW, Lu CF, Chang ST, Tsai PY. Functional Near-Infrared Spectroscopy as a Target Navigator for rTMS Modulation in Patients with Hemiplegia: A Randomized Control Study. Neurol Ther. 2022 Mar;11(1):103-121. doi: 10.1007/s40120-021-00300-0. Epub 2021 Nov 13. PMID 34773596
- [Derived] Tsai PY, Lin WS, Tsai KT, Kuo CY, Lin PH. High-frequency versus theta burst transcranial magnetic stimulation for the treatment of poststroke cognitive impairment in humans. J Psychiatry Neurosci. 2020 Jul 1;45(4):262-270. doi: 10.1503/jpn.190060. PMID 32159313
- [Derived] Lai CJ, Wang CP, Tsai PY, Chan RC, Lin SH, Lin FG, Hsieh CY. Corticospinal integrity and motor impairment predict outcomes after excitatory repetitive transcranial magnetic stimulation: a preliminary study. Arch Phys Med Rehabil. 2015 Jan;96(1):69-75. doi: 10.1016/j.apmr.2014.08.014. Epub 2014 Sep 11. PMID 25218256
- See also: Document of rTMS effect in functional facilitation — http://www.ncbi.nlm.nih.gov/pubmed/23194830
- See also: Document of rTMS effect in functional facilitation — http://www.ncbi.nlm.nih.gov/pubmed/21980359
- See also: Document of rTMS effect in functional facilitation — http://www.ncbi.nlm.nih.gov/pubmed/19309294